CLINICAL TRIAL: NCT04341922
Title: Evaluation of a Brief Online-delivered Cognitive-behavioral Intervention for Dysfunctional Worry Related to the Covid-19 Pandemic: A Randomized Controlled Trial
Brief Title: A Online-delivered Cognitive-behavioral Intervention for Dysfunctional Worry Related to the Covid-19 Pandemic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erik Andersson, PhD, psychologist, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2020-01719
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Dysfunctional Worry
Keywords: Covid-19; internet-delivered; cognitive behavioral intervention
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Online Cognitive-Behavioral intervention (Experimental): The three-week intervention is a structured self-guided program without therapist support, administered via a secure web platform and organized in five brief modules. The treatment is provided through an encrypted online platform (login through BankID and double authentication) provided by the eHealth Core facility at Karolinska Institutet
  Interventions: Behavioral: Internet-delivered cognitive behavior therapy (ICBT) for dysfunctional worry related to the Covid-19 pandemic
- Wait-list (No Intervention): The wait-list controlled composes of no intervention for three weeks. Participants randomized to the wait-list group will be crossed over to receive the Online Cognitive-Behavioral intervention after three weeks (post-treatment).

INTERVENTIONS:
Behavioral: Internet-delivered cognitive behavior therapy (ICBT) for dysfunctional worry related to the Covid-19 pandemic — The intervention focuses on 1) teaching participants how to discriminate between functional and dysfunctional worry (what are solvable problems vs. what is worry, i.e. unsolvable thoughts?) 2) providing participants with skills to solve functional worry topics (e.g. set time and make a workable plan to be prepared for possible negative outcomes [e.g. becoming unemployed]), 3) helping participants to reduce unhelpful behaviors that may reinforce worry (e.g., limit excessive news consumption, refrain from assurance seeking behaviors), 4) providing participants with skills to approach dysfunctional worry (e.g., not engage in worrisome thoughts, just leave them), and 5) increase the behavioral repertoire (take walks, engage in activities that promote health without putting oneself at risk to become infected).
  Arms: Intervention: Online Cognitive-Behavioral intervention

SUMMARY:
The purpose of this study is to investigate if a brief online-delivered cognitive-behavioral intervention can reduce the degree of dysfunctional worry related to the Covid-19 pandemic, compared to a wait-list control condition.

DETAILED DESCRIPTION:
Worries about the immediate and long-term consequences of the ongoing Covid-19 pandemic are largely justified in the current climate of uncertainty. However, dysfunctional worry, that is, pervasive worry that is disproportionate in its intensity or duration, and that significantly interferes with every-day problem-solving or goal-driven behavior, is clearly counterproductive. Research has also indicated that repeated media exposure to a community crisis can lead to increased anxiety and heightened stress responses, that can give a downstream effect on health, and misplaced health-protective and help-seeking behaviors which, in turn, may overburden health care facilities. There is an urgent need to develop a brief, scalable intervention to target such dysfunctional worry in the general population.

The current randomized controlled trial will evaluate the feasibility and efficacy of a brief online-delivered cognitive behavioral intervention designed to target dysfunctional worry related to the Covid-19 pandemic. 670 individuals are randomized to intervention or to waiting-list. The hypothesis is that the brief self-guided intervention will show significant within-group reductions in self-rated worry from baseline (week 0) to post-treatment (week 3), and that these improvements will be larger than those seen in the wait-list control group. The wait-list group will be crossed over to receive the intervention after three weeks (post-treatment). All participants will be followed-up one month and one year after the end of the intervention.

ELIGIBILITY:
INCLUSION CRITERIA

* The following 2 criteria must be met:

  * Worrying about Covid-19 and its possible consequences (e.g. risk of getting ill, fear of death, economy, family, etc.) every day, often several times a day
  * The worry about Covid-19 is perceived as difficult to control
* In addition, at least one of the following negative consequences of worrying:

  * The worry about Covid-19 takes so much time and energy that it is difficult to concentrate on anything else (work, family, hobbies, etc.)
  * Trouble sleeping due to Covid-19 worries
  * Constantly checking the news and social media to follow developments about Covid-19
  * Marked loss of work productivity due to worries about Covid-19
  * Difficulties finding joy in everyday situations because of worry about Covid-19
* ≥ 18 years of age
* Resident in Sweden
* Daily access to a computer or other device with internet connection

EXCLUSION CRITERIA

* Non Swedish speaking
* Severe depression, defined as >28 points on the MADRS-S
* Suicidal risk defined as 5 points or above on item 9 on the MADRS-S
* Family member in the same household who is included in the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 670 (Actual)
Dates: Start 2020-05-09 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2021-09-10 (Estimated)

PRIMARY OUTCOMES:
• Covid-19-adapted version of the self-rated Generalized Anxiety Disorder Scale-7 (GAD-7) | Basline (week 0), during treatment (week 1 and week 2), post treatment (week 3), at one-month after treatment and also one year follow up.
  A 7-item self-rated scale to assess symtom severity of worry. Total score ranging from 0 to 21. Effects will be expressed as the change from baseline to last post-treatment value (Week 0-Week 3) period. Effects will also be assessed at one month and one year post-treatment.

SECONDARY OUTCOMES:
Montgomery Åsberg Depression Rating Scale - Self report (MADRS-S) | Baseline (week 0), post treatment (week 3), at one-month after treatment and also one year follow up.
  A 9-item self-rated scale to assess symtoms of depression.Total score ranging from 0 to 54.
Adapted Covid-19 version of the Work and Social Adjustment Scale (WSAS) | Basline (week 0), during treatment (week 1 and week 2), post treatment (week 3), at one-month after treatment and also one year follow up.
  A 5-item self-rated scale adapted to measure impact of the Covid-19 pandemic on work and social functioning. Total score ranging from 0 to 40.
Insomnia Severity Index (ISI) | Baseline (week 0), post treatment (week 3), at one-month after treatment and also one year follow up.
  A 7-item self-rated scale to asess severity of insomnia symtoms. Total score ranging from 0 to 28.
Adapted Swedish version of the CoRonavIruS Health Impact Survey (CRISIS) | Baseline (week 0), post treatment (week 3), at one-month after treatment and also one year follow up.
  A self-rated scale to assess Coronavirus/covid-19 health/exposure status, life changes, changes in daily behaviors, impact on emotions/worries, changes in media use past two weeks and changes in substance use due to coronavirus/covid-19 crisis. The scale has bees translated to Swedish and adopted to a Swedish context.
Intolerance of uncertainty Scale (IUS) | Baseline (week 0), post treatment (week 3), at one-month after treatment and also one year follow up.
  A 12-item self-rated scale to assess intolerance of uncertainty. Total score ranging from 12 to 60.
Patient Satisfaction Questionnaire (PSQ) | Post treatment (week 3)
  A self-rated scale to assess treamtent satisfaction.
Adverse events (AE) | Post treatment (week 3)
  A self-rated questionnaire with free text options to assess adverse events du to the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Erik M Andersson, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Derived] Wahlund T, Mataix-Cols D, Olofsdotter Lauri K, de Schipper E, Ljotsson B, Aspvall K, Andersson E. Brief Online Cognitive Behavioural Intervention for Dysfunctional Worry Related to the COVID-19 Pandemic: A Randomised Controlled Trial. Psychother Psychosom. 2021;90(3):191-199. doi: 10.1159/000512843. Epub 2020 Nov 19. PMID 33212440